CLINICAL TRIAL: NCT02526966
Title: Multicenter Study Evaluating the Performance of the Assay of Anti-hinge Region Antibodies in the Diagnosis of Progressive Forms of IgA Nephropathy
Acronym: NIGA-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1108060; 2011-A00860-41 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-03

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with primitive form of IgA nephropathy (Other)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — dosage of anti-hinge region antibodies

SUMMARY:
The anti-hinge region antibodies would be a relevant biomarker of IgA nephropathy. Beyond a prognostic value (which could increase the risk of Renal Absolute), the longitudinal monitoring for these antibodies could be of interest: (1) in the monitoring of patients (in place including a possible repetition renal biopsy); (2) to guide treatment decisions and (3) in clinical research, as an outcome (in substitution for the occurrence of kidney failure) in therapeutic trials IgA nephropathy.

This research project constitutes the first step in validating these antibodies biomarker of IgA nephropathy and its main objective is to study the performance of the blood levels of anti-hinge region antibodies in the diagnosis of progressive forms of histologically IgA nephropathy as defined by the Renal Risk Absolute.

The secondary objectives of this project are to establish a bio-collection that will allow us to search for other prognostic factors (genetic, cellular and serum) of IgA nephropathy and to evaluate the performance of Renal Absolute risk by integrating Oxford score, the new international histological classification.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient
* Diagnosis of a primitive form of IgA nephropathy histologically proven

Exclusion Criteria:

* Suspicion of secondary IgA nephropathy forms
* Less than 5 glomeruli present on renal biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
serum concentration of anti-hinge region antibodies (mg/ml) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MARIAT, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (15):
- France (15):
  - CH d'ANNECY, Annecy
  - CH d'ANNONAY, Annonay
  - CH de BOURG EN BRESSE, Bourg-en-Bresse
  - CH de CHAMBERY, Chambéry
  - CHU de CLERMONT-FERRAND, Clermont-Ferrand
  - CHU de DIJON, Dijon
  - CHU de GRENOBLE, Grenoble
  - CH du PUY EN VELAY, Le Puy-en-Velay
  - Hôpital Edouard. HERRIOT, Lyon
  - Centre Hospitalier de Lyon Sud, Pierre-Bénite
  - CH de ROANNE, Roanne
  - Hôpitaux Drome Nord, Romans
  - CHU de SAINT-ETIENNE, Saint-Etienne
  - CH de VALENCE, Valence
  - Clinique du TONKIN, Villeurbanne

IPD SHARING:
Plan to Share IPD: No